CLINICAL TRIAL: NCT03577106
Title: A Pilot fMRI Study of TMS in Late-Life Severe Worry
Acronym: TINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmen Andreescu (Other)
Responsible Party: Sponsor-Investigator, Carmen Andreescu, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19020109
Record Dates: First submitted 2018-05-31; First posted 2018-07-05 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Anxiety Disorders Generalized
Keywords: transcranial magnetic stimulation; TMS; MRI; magnetic resonance imaging; fMRI; functional magnetic resonance imaging; sleep; intermittent theta burst stimulation; iTBS
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Transcranial magnetic stimulation (TMS) (Experimental)
  Interventions: Device: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Device: Transcranial magnetic stimulation (TMS) — Theta Burst Stimulation (TBS), a form of TMS, will be targeted to the Inferior Parietal Cortex based on neural navigation software. TBS will be delivered for about 5-6 minutes, five days a week for two weeks, for a total of ten sessions.

SUMMARY:
Investigators will test a novel intervention through experimental therapeutic approach using fMRI-directed Intermittent Theta Burst Stimulation (iTBS), a high frequency TMS paradigm, for the treatment of severe, uncontrollable worry. While worry is a universal human experience, severe and excessive worry has been recently linked to increased risk of stroke and other cardiovascular diseases, increased risk of conversion to Alzheimer's disease as well as to higher risk of all-cause mortality in midlife and late-life. Severe, uncontrollable worry has been repeatedly associated with reduced quality of life and impaired functioning. Current treatment choices (antidepressant/anxiolytic medications and psychotherapeutic interventions) have been proven moderately efficacious in reducing anxiety/depression burden, but ineffective in reducing worry severity, a phenomenon that may contribute to the high relapse rates associated with mood and anxiety disorders. Our research indicated that worry severity is associated with hyperactivation in specific regions such as orbital frontal cortex, superior parietal gyrus, amygdala and parahippocampal gyrus. This pilot study will explore the efficacy of targeting one of these regions with iTBS. Based on investigators' previous results, the most accessible target is the right superior parietal gyrus (rSPG) - a region that remained significantly associated with severe worry after controlling for effects of comorbid depression or overall anxiety. As this region showed an increased in cerebrovascular flow in association with worry severity, investigators will use iTBS (5x/week for 2 weeks) to modulate cortical plasticity in this region and consequently, to reduce worry severity.

TMS during wakefulness has been shown to alter subsequent sleep [4], Further, changes in sleep in response to TMS has been associated with how participants respond to the TMS as a treatment [5]. Thus, the study will measure sleep throughout the protocol to determine whether sleep changes as a function of TMS and whether sleep changes are associated with treatment response.

DETAILED DESCRIPTION:
Background:

Twenty percent of older adults in the community report severe worry. While worry is a universal human experience, severe and excessive worry in older adults has been recently linked to increased risk of stroke and other cardiovascular diseases, increased risk of conversion to Alzheimer's disease as well as to higher risk of all-cause mortality. As worry is a transdiagnostic construct, it is present in several mood and anxiety disorders, including major depressive disorder and generalized anxiety disorder. Current treatment choices in late-life (antidepressant/anxiolytic medications and psychotherapeutic interventions) have been proven moderately efficacious in reducing anxiety/depression burden, but ineffective in reducing worry severity, a phenomenon that may contribute to the high relapse rates associated with mood and anxiety disorders in the geriatric population. These elements support the need for novel, experimental interventions specifically designed to target the neural basis of severe worry in late-life. Through a pre-existing study (R01 MH108509), investigators focus on describing the behavior of canonical neural networks during resting state and during worry induction in participants with low-to-high worry. The research indicates that simple induction of worry activates a distinct set of regions (caudate/thalamus, visual cortex, dorsal anterior cingulate). Given the universality and potential evolutionary benefits of worry, investigators believe that the neural network associated with worry induction supports a normal, physiologic experience. However, the regions involved in maintaining worry (hippocampus, thalamus) as well as those associated with severe worry (orbitofrontal cortex, superior parietal gyrus, amygdala, parahippocampal gyrus) support a pathological phenomenon and may represent ideal targets for interventions.

This pilot study will test the engagement of therapeutic targets during TBS. Based on the investigators' preliminary results, the most accessible and relevant target is the parietal cortex - a region that in the investigators K 23 sample remained significantly associated with severe worry after controlling for effects of comorbid depression or overall anxiety. As parietal cortex cerebrovascular flow increased in association with worry severity, the investigators will use inhibitory TBS [high frequency TMS at 1 Hz] to modulate cortical plasticity and consequently reduce worry severity. To test target engagement, the research team will use the in-scanner worry induction paradigm designed by Dr. Andreescu and her mentors during her K23 award and currently use to probe worry induction in the R01 MH108509. Given the exploratory nature of this proposal and based on our preliminary data, we will use two measures of target engagement: 1) the relative decrease in BOLD signal in the parietal cortex and 2) the relative decrease in rSPG-dACC functional connectivity.

Significance:

1. Severe worry in late-life carries a significant health care risk. Worry is defined as a complex affective and cognitive process, negative-affect laden, and relatively uncontrollable [6]. While worry is a universal human experience that may confer an evolutionary advantage by modifying threat-related decision-making, severe and excessive worry has been recently linked to increased risk of conversion from mild cognitive impairment to Alzheimer's disease [7], and with increased risk of stroke and other cardiovascular events, after controlling for depression and vascular risk factors. Severe worry is also associated with interruption in functioning and reduced quality of life and with a higher risk of all-cause mortality in midlife and late-life.
2. Severe worry in late-life responds poorly to traditional interventions. Traditionally, severe worry has been confined to categories such as Generalized Anxiety Disorder (GAD) and Major Depressive Disorder (MDD), multiple lines of research support the presence of severe worry in other several other anxiety and mood disorders. Thus, while GAD is built around the concept of severe, uncontrollable worry, only 20% of severe older worriers qualify for a GAD diagnosis. This evidence supports a major recent shift in the conceptualization of worry as a transdiagnostic entity most suitable for dimensional investigations. Current late-life GAD treatment choices, including cognitive-behavioral therapy (CBT) and antidepressant pharmacotherapy, have proven moderately efficacious in reducing overall burden of anxiety but ineffective in reducing worry severity. The ineffectiveness of current treatments in reducing worry severity may be at the root of the chronic, relapsing course of late-life GAD, which is one of the least likely mental disorders to remit and most likely to relapse.
3. Novel circuit-based targets for intervention. Several neuroimaging studies have investigated both activation and functional connectivity among various brain regions involved in GAD - in adolescents and young adults. This research team has published exclusively on the neural markers of GAD in older adult participants. Also, very few studies used fMRI paradigms specifically tailored to induce worry or analyzed specifically the effect of worry severity at rest or during task. The investigators' current results point toward two different networks that may benefit from targeted interventions: the one associated exclusively with severe worry (amygdala-parahippocampus- rOFC- rSPG) and the one associated with maintenance/the protracted quality of worry (insula-caudate/thalamus-amygdala-parahippocampus).

The investigators decided to target the network associated with worry severity due to both the richer literature regarding the pernicious effect of severe worry on both public health and treatment response but also due to accessibility for TMS of the rSPG. Overall, the worry severity network seems to implicate excessive limbic/paralimbic activation potentially amplified by the cognitive anticipation of the negative affective value of future events processed through the OFC as well as probable attempts to cognitively control the arousal and dysphoria through structures such as dACC and SPG. This speculation is in line with newer interpretations of pathologic worry that suggest severe worriers both maintain arousal in order to seek out potential solutions to the anxiogenic source while attempting to inhibit representations of the potential bad outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have completed Dr. Andreescu's study R01MH108509/PRO15080120.
* Penn State Worry Questionnaire score of 55 or above.

Exclusion Criteria:

* Any form of psychosis or Bipolar Disorder, dementia, a history of substance abuse within the last six months
* Use of antidepressants within the last five to fourteen days (adequate washout interval to be determined by the principal investigator (PI) based on each specific antidepressant). For fluoxetine, the washout interval will be six weeks. However, for participants who are prescribed low dose psychotropics for pain, sleep disturbances, and/or medical conditions (e.g. amitriptyline for peripheral neuropathy, low dose trazodone as a sleep aid), these will be allowed in most circumstances. We will include participants on certain dosages of the most commonly prescribed antidepressants (for medical reasons) as follows: amitriptyline up to 50 mg/d, doxepin up to 50 mg/d, trazodone up to 100 mg/d, and imipramine up to 50 mg/d. We will review other cases individually and the PI will decide if the participants are eligible for the study and if they may continue the current medication.
* Unable to complete MRI scans: presence of ferromagnetic metal in the body, claustrophobia
* Contraindications for TMS:

  1. Presence of a neurologic disorder or medical condition known to alter seizure threshold(e.g., stroke, aneurysm, brain surgery, structural brain lesion, brain injury, frequent/severe headaches)
  2. Recurrent seizures or epilepsy in participant
  3. Pregnancy
  4. Metallic implants in body located at 30 cm or less from the position of the magnetic coil; presence in the body of other devices that may be affected by magnetic field (e.g. pacemakers).
* Unable to temporarily discontinue benzodiazepines 48 hours prior to MRI scan. Participants on high doses of benzodiazepines (e.g., greater than or equivalent to 2 mg of lorazepam) will be excluded, given the complexity and potential complications of benzodiazepine taper/withdrawal.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Andreescu, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saeki T, Nakamura M, Hirai N, Noda Y, Hayasaka S, Iwanari H, Hirayasu Y. Localized potentiation of sleep slow-wave activity induced by prefrontal repetitive transcranial magnetic stimulation in patients with a major depressive episode. Brain Stimul. 2013 May;6(3):390-6. doi: 10.1016/j.brs.2012.08.004. Epub 2012 Aug 31. PMID 22964349
- [Background] Rosenquist PB, Krystal A, Heart KL, Demitrack MA, McCall WV. Left dorsolateral prefrontal transcranial magnetic stimulation (TMS): sleep factor changes during treatment in patients with pharmacoresistant major depressive disorder. Psychiatry Res. 2013 Jan 30;205(1-2):67-73. doi: 10.1016/j.psychres.2012.09.011. Epub 2012 Sep 25. PMID 23021320
- [Background] Golden J, Conroy RM, Bruce I, Denihan A, Greene E, Kirby M, Lawlor BA. The spectrum of worry in the community-dwelling elderly. Aging Ment Health. 2011 Nov;15(8):985-94. doi: 10.1080/13607863.2011.583621. Epub 2011 Jul 12. PMID 21749221
- [Background] Tully PJ, Cosh SM, Baune BT. A review of the affects of worry and generalized anxiety disorder upon cardiovascular health and coronary heart disease. Psychol Health Med. 2013;18(6):627-44. doi: 10.1080/13548506.2012.749355. Epub 2013 Jan 16. PMID 23324073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 63 participants from the parent study, FINA, were phone screened for this study. 28 of those individuals signed consent for this study, but 4 of the 28 were deemed ineligible for the study prior to the TMS intervention, leaving a total of 24 participants being enrolled in the study that received at least 1 session of TMS treatment.
Pre-assignment Details: After signing consent, but prior to starting the TMS intervention, participants were asked to complete a Penn State Worry Questionnaire to assess anxiety/worry levels. Individuals with a PSWQ score of 55 or higher qualified for the study intervention, and those with a score of 54 or lower were excluded from the study. Participants with low PSWQ scores were excluded as treatment was relevant only for high worriers.
Period: Overall Study
Arm/Group | Transcranial Magnetic Stimulation (TMS)
Started | 24
Completed | 21
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Number of participants who started at least 1 session of TMS provided by the study
Arm/Group | Transcranial Magnetic Stimulation (TMS)
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 19
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
Penn State Worry Questionnaire (PSWQ) Score [Mean (Full Range); unit: units on a scale] — PSWQ scores can range from 16 to 80, where a lower score represents a better outcome of having lower levels of worry. Population: PSWQ analysis includes only the 21 participants who completed the full trial of TMS treatment. The 3 participants who withdrew from the study were not included within this data as they do not have follow-up PSWQ scores to analyze.
  units on a scale
    number analyzed (Participants) | 21
    (all) | 68.62 [58 to 80]

OUTCOME MEASURES:

1. Primary Outcome: Change in Worry Severity From Baseline to Post-intervention as Measured by the Penn State Worry Questionnaire (PSWQ)
Description: Penn State Worry Questionnaire (PSWQ) scores range from 16 to 80 with higher levels indicating greater worry severity.
Time Frame: Baseline and within 2 weeks post-TMS intervention
Population: Participants who completed study TMS protocol
Measure: Mean (Standard Deviation); unit: units on a scale (PSWQ)
Arm/Group | Transcranial Magnetic Stimulation (TMS)
Number analyzed (Participants) | 21
units on a scale (PSWQ)
  PSWQ Score after TMS Treatment | 62.43 (10.28)
  Change from Baseline at Two Weeks | 6.19 (8.5)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation (TMS); Mean difference using a paired t-test; Test type: Other; p < 0.005, paired t-test — t(20)=3.3, p<0.005

2. Primary Outcome: Participants Who Responded to TMS
Description: The breakdown of participants who responded to TMS treatment; responders had Penn State Worry Questionnaire (PSWQ) scores that decreased by 30% or more from the baseline timepoint to the end of TMS treatment.
Time Frame: Baseline and the end of TMS intervention (approximately two weeks)
Population: The breakdown of participants who responded to TMS treatment; responders had Penn State Worry Questionnaire (PSWQ) scores that decreased by 30% or more from the baseline timepoint to the end of TMS treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Transcranial Magnetic Stimulation (TMS)
Number analyzed (Participants) | 21
Participants
  TMS Responders | 2
  TMS Non-responders | 19

ADVERSE EVENTS:
Time Frame: Adverse events were systematically assessed daily for the 2 weeks of TMS treatment for each participant, and non-systematically assessed as needed throughout the entire study, an average of 6 weeks.
Description: Participants were monitored throughout the TMS protocol, and asked twice a session to describe any discomfort they experienced, along with rating this discomfort on a scale. Participants were also able to report discomfort at any time during treatment, to which the study team would respond accordingly.
Arm/Group | Transcranial Magnetic Stimulation (TMS)
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 1/24
Other Adverse Events (participants affected / at risk) | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial Magnetic Stimulation (TMS) (N=24)
Kidney Stone (Renal and urinary disorders) | 1 (1) — One participant experienced having a kidney stone during the course of their TMS treatment within the study. They were hospitalized for this, and missed the final TMS session. This was not related to study intervention but was unanticipated.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Transcranial Magnetic Stimulation (TMS) (N=24)
Jaw clenching/Teeth Rattling (Musculoskeletal and connective tissue disorders) | 20 — The stimulation from the TMS coil can also activate the jaw muscles, which can result in participants clenching their jaw or having their teeth rattle. This event was expected, and was mediated with putting gauze in participant's mouths beforehand.
Tapping Sensation on Scalp/Eye or Cheek Twitch (Skin and subcutaneous tissue disorders) | 21 — Activation of the neurons within the brain via the TMS coil also creates a tapping sensation on the scalp for the person receiving treatment. This can also translate across the face to make the eye or cheek twitch. This event was anticipated.
Neck Muscle Twitching (Musculoskeletal and connective tissue disorders) | 2 — TMS stimulation may also cause participant's neck muscles to twitch, similar to having jaw muscles twitch. This event was anticipated.
Headache (Musculoskeletal and connective tissue disorders) | 9 — TMS stimulation can cause headaches at the site of treatment during or immediately after treatment. These headaches are usually reported as being either tension headaches, or as feeling like a dull ache. Headaches were an anticipated event.
Unsteadiness/Dizziness (General disorders) | 3 — Some participants experienced a brief degree of unsteadiness or dizziness upon exiting the TMS treatment chair.

LIMITATIONS AND CAVEATS:
Due to COVID, we were only able to recruit a total of 21 participants instead of 40 who were to complete full treatment. The treatment was only a typical 'half' dose consisting of 10 sessions of TMS rather than 20, which is typical. Three participants started TMS and decided to withdraw due to discomfort from TMS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT03577106/Prot_SAP_003.pdf